CLINICAL TRIAL: NCT05503602
Title: Investigation of the Effect of Instrument Assisted Soft Tissue Mobilization Technique and Foam Roller Application on Strength, Flexibility, Pain and Secondary Outcome Measures in Individuals With Chronic Non-Specific Neck Pain.
Brief Title: Investigation of the Effect of Instrument Assisted Soft Tissue Mobilization Technique and Foam Roller Application in Individuals With Chronic Non-Specific Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Muhammed Usame TAS, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ÜSAME TAŞ-001
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Instrument-assisted Soft Tissue Mobilization; Flexibility; Foam Roller; Strength; Chronic Non-specific Neck Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Other): An average of 20 people will be taken into the control group.
  Interventions: Other: Classical Physiotherapy
- IASTM Treatment Group (Experimental): An average of 20 people will receive IASTM application treatment.
  Interventions: Other: IASTM Technique Application
- Foam Roller Treatment Group (Experimental): An average of 20 people will receive Foam Roller application treatment.
  Interventions: Other: Foam Roller Technique Application

INTERVENTIONS:
Other: Classical Physiotherapy — Only classical physiotherapy application, 5 sessions per week for 4 weeks.
  Arms: Control Group
Other: IASTM Technique Application — Instrument-assisted soft tissue mobilization application 2 sessions per week together with 3 sessions of classical physiotherapy per week for 4 weeks. IASTM application; A total of 4 minutes will be applied to the sternocleidomastoideus, levator scapula, scalene muscles and upper part of the trapezius for a total of 4 minutes (2 minutes to the right, 2 minutes to the left region).
  Arms: IASTM Treatment Group
Other: Foam Roller Technique Application — 2 sessions of foam roller technique per week along with 3 sessions of classical physiotherapy per week for 4 weeks. Foam roller application; A total of 4 minutes will be applied to the sternocleidomastoideus, levator scapula, scalene muscles and upper part of the trapezius for a total of 4 minutes (2 minutes to the right, 2 minutes to the left region).
  Arms: Foam Roller Treatment Group

SUMMARY:
Neck pain is in fourth place among the pathologies that result in the state of disability. Acute neck pain improves greatly within 2 months, while neck pain that persists for more than 3 months takes the form of chronic neck pain. Pain adversely affects people's activities of daily living. Treatment applications such as electrotherapy, hot and cold applications are applied for purposes such as reducing pain and muscle spasm and correcting functions. In addition to such treatment options, instrument-assisted soft tissue mobilization (IASTM) and foam roller therapy have been started to be applied in many disease groups in recent years and have attracted great attention. iASTM and Foam Roller is a technique that involves the use of tools in disorders of musculoskeletal pathology and to help heal soft tissues.

The aim of this study is to investigate the effects of foam roller technique with instrument-assisted soft tissue mobilization technique in individuals of different ages with chronic non-specific neck pain. According to the data obtained, the techniques the investigators will use, together with physiotherapy programs, contribute to the treatment of individuals with chronic non-specific neck pain and to the literature.is expected to provide.

DETAILED DESCRIPTION:
In the study, Foam Roller will be applied to individuals with chronic non-specific neck pain with iASTM and the effect of these techniques will be examined. Demographic information of individuals will be recorded; individuals will be evaluated in detail in terms of muscle strength, flexibility, pain and secondary outcome measures. Individuals in terms of secondary outcome measures; functional status,joint range of motion and quality of life will be evaluated.

The work plan; pre-treatment evaluation, followed by treatment, second evaluation immediately after the end of treatment and control evaluation (third evaluation) 1 month after the end of treatment. The data collection period is planned as 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Consists of individuals between the ages of 18-60,
2. Being diagnosed with chronic non-specific neck pain,
3. Having a score of at least 4 on the visual analog scale (VAS) of the mean neck pain intensity,
4. Having non-specific neck pain at least 5 days a week for the last 12 weeks,
5. To be deemed appropriate by the physical therapy physician for early physiotherapy treatment after the diagnosis of chronic non-specific neck pain.

Exclusion Criteria:

1. Individuals with a history of cervical spine surgery, cervical trauma, central nervous system diseases, cervical radiculopathy, acute inflammation and malignancy,
2. Having neck pain due to specific causes (disc protrusion, radicular syndrome, whiplash, congenital deformity of the spine, spinal canal stenosis and neoplasm),
3. Individuals with inflammatory rheumatic disease, active oncological disease, affective disorder, addiction and psychosis,
4. Individuals who have undergone invasive treatment of the spine in the last 4 weeks or spine surgery in the previous 12 months,
5. Individuals from the chronic neck pain group who are currently receiving treatment or have a neck injury resulting in a spinal fracture,
6. Individuals who have started a new treatment for neck pain in the past month or are planning to start a new treatment within 9 weeks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Muscle Strength Assessment | Pre-treatment assessment.
  A digital muscle dynamometer will be used to evaluate the muscle strength of the patients.
Muscle Strength Assessment | Second evaluation immediately after the end of 4 weeks of treatment.
  A digital muscle dynamometer will be used to evaluate the muscle strength of the patients.
Muscle Strength Assessment | Control evaluation 1 month after the end of treatment (third evaluation).
  A digital muscle dynamometer will be used to evaluate the muscle strength of the patients.
Flexibility Assessment | Pre-treatment assessment.
  A tape measure will be used to assess patients' flexibility. The ear-shoulder, chin-sternum (proximal end) and chin-wall distances of the patients will be measured with a tape measure.
Flexibility Assessment | Second evaluation immediately after the end of 4 weeks of treatment.
  A tape measure will be used to assess patients' flexibility. The ear-shoulder, chin-sternum (proximal end) and chin-wall distances of the patients will be measured with a tape measure.
Flexibility Assessment | Control evaluation 1 month after the end of treatment (third evaluation).
  A tape measure will be used to assess patients' flexibility. The ear-shoulder, chin-sternum (proximal end) and chin-wall distances of the patients will be measured with a tape measure.
Pain Assessment | Pre-treatment assessment.
  Visual Analog Scale (VAS) will be used to evaluate the pain of individuals.
Pain Assessment | Second evaluation immediately after the end of 4 weeks of treatment.
  Visual Analog Scale (VAS) will be used to evaluate the pain of individuals.
Pain Assessment | Control evaluation 1 month after the end of treatment (third evaluation).
  Visual Analog Scale (VAS) will be used to evaluate the pain of individuals.

SECONDARY OUTCOMES:
Functional Status Assessment Questionnaire | Pre-treatment assessment.
  Neck Disability Index (NDI) will be used to evaluate the functional status of patients. The NDI consists of 10 titles: pain severity, self-care, lifting, reading, headache, concentration, working, driving, sleeping and recreation. Individuals included in the study are asked to give points between 0 (no disability) and 5 (complete disability) to each title. The total score ranges from 0 (no disability) to 50 (complete disability).
Functional Status Assessment Questionnaire | Second evaluation immediately after the end of 4 weeks of treatment.
  Neck Disability Index (NDI) will be used to evaluate the functional status of patients. The NDI consists of 10 titles: pain severity, self-care, lifting, reading, headache, concentration, working, driving, sleeping and recreation. Individuals included in the study are asked to give points between 0 (no disability) and 5 (complete disability) to each title. The total score ranges from 0 (no disability) to 50 (complete disability).
Functional Status Assessment Questionnaire | Control evaluation 1 month after the end of treatment (third evaluation).
  Neck Disability Index (NDI) will be used to evaluate the functional status of patients. The NDI consists of 10 titles: pain severity, self-care, lifting, reading, headache, concentration, working, driving, sleeping and recreation. Individuals included in the study are asked to give points between 0 (no disability) and 5 (complete disability) to each title. The total score ranges from 0 (no disability) to 50 (complete disability).
Joint Range of Motion Assessment | Pre-treatment assessment.
  A goniometer will be used to evaluate the patients' range of motion.
Joint Range of Motion Assessment | Second evaluation immediately after the end of 4 weeks of treatment.
  A goniometer will be used to evaluate the patients' range of motion.
Joint Range of Motion Assessment | Control evaluation 1 month after the end of treatment (third evaluation).
  A goniometer will be used to evaluate the patients' range of motion.
Quality of Life Assessment Questionnaire | Pre-treatment assessment.
  The Nottingham Health Profile (NHP) will be used to assess patients' quality of life. The Nottingham health profile is a scale used to assess patients' levels of emotional, social and physical activity. The questions are divided into 6 subgroups as energy level (3 questions), pain (8 questions), emotional reaction (9 questions), sleep (5 questions), social isolation (5 questions) and physical activity limitation (8 questions). A total of 38 questions in 6 groups have separate point values, and each item is answered "yes" or "no". A scoring system has been established so that each subgroup will have a total of 100 points.
Quality of Life Assessment Questionnaire | Second evaluation immediately after the end of 4 weeks of treatment.
  The Nottingham Health Profile (NHP) will be used to assess patients' quality of life. The Nottingham health profile is a scale used to assess patients' levels of emotional, social and physical activity. The questions are divided into 6 subgroups as energy level (3 questions), pain (8 questions), emotional reaction (9 questions), sleep (5 questions), social isolation (5 questions) and physical activity limitation (8 questions). A total of 38 questions in 6 groups have separate point values, and each item is answered "yes" or "no". A scoring system has been established so that each subgroup will have a total of 100 points.
Quality of Life Assessment Questionnaire | Control evaluation 1 month after the end of treatment (third evaluation).
  The Nottingham Health Profile (NHP) will be used to assess patients' quality of life. The Nottingham health profile is a scale used to assess patients' levels of emotional, social and physical activity. The questions are divided into 6 subgroups as energy level (3 questions), pain (8 questions), emotional reaction (9 questions), sleep (5 questions), social isolation (5 questions) and physical activity limitation (8 questions). A total of 38 questions in 6 groups have separate point values, and each item is answered "yes" or "no". A scoring system has been established so that each subgroup will have a total of 100 points.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Üsame TAŞ, Lecturer, Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No